CLINICAL TRIAL: NCT03620747
Title: Open-label, Interventional, Cohort Study to Evaluate Long-term Safety of Dupilumab in Patients With Moderate to Severe Asthma Who Completed the TRAVERSE-LTS12551 Clinical Trial
Brief Title: Continuation of TRAVERSE- LTS12551 Evaluating Dupilumab Safety in Patients With Asthma (Long-Term Follow-Up)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS15023; 2017-002134-23 (EudraCT Number); U1111-1196-5369 (Other: UTN)
Record Dates: First submitted 2018-07-26; First posted 2018-08-08 (Actual); Results first posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dupilumab (Experimental): Participants received subcutaneous (SC) dose of dupilumab 300 milligrams (mg) every 2 weeks (q2w) from Week 0 up to Week 132. Participants who discontinued treatment for greater than or equal to (>=) 6 weeks after study LTS12551 (NCT02134028), received a 600 mg loading dose of dupilumab on Week 0. Participants were also on background dose of medium or high dose inhaled corticosteroid (ICS) as maintained in study LTS12551 in combination with controllers (and/or oral corticosteroid [OCS] for those participants from the original parent study EFC13691 [NCT02528214]). Salbutamol/albuterol hydrofluoroalkane pressurized metered dose inhalers (MDI) or levosalbutamol/levalbuterol hydrofluoroalkane pressurized MDI were given as reliever medication as needed during the study.
  Interventions: Drug: Dupilumab SAR231893 (REGN668)

INTERVENTIONS:
Drug: Dupilumab SAR231893 (REGN668) — Pharmaceutical form: prefilled syringes
  Route of administration: subcutaneous

SUMMARY:
Primary Objective:

To describe the long-term safety of dupilumab in treatment of participants with moderate to severe asthma who completed the previous asthma clinical trial (TRAVERSE-LTS12551).

DETAILED DESCRIPTION:
Duration per participant was until dupilumab approval for use in asthma and market availability to the participant, or a maximum of 144 weeks (i.e., about 3 years) after the start of treatment (Visit 1), whichever came first.

ELIGIBILITY:
Inclusion criteria:

* Participants with asthma who completed the treatment period in the previous dupilumab asthma clinical study LTS12551.
* Signed written informed consent.

Exclusion criteria:

* Participants who experienced any systemic hypersensitivity reactions to the investigational medicinal product in the previous dupilumab asthma study LTS12551, which, in the opinion of the Investigator, could indicate that continued treatment with dupilumab might present an unreasonable risk for the participant.
* Clinically significant comorbidity/lung disease other than asthma.
* Participants with active autoimmune disease or participants who, as per Investigator's medical judgment, were suspected of having high risk for developing autoimmune disease.
* History of malignancy within 5 years before enrollment except completely treated in situ carcinoma of the cervix, completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (132):
- United States (35):
  - Investigational Site Number :840099, Gilbert, Arizona
  - Investigational Site Number :840087, Scottsdale, Arizona
  - Investigational Site Number :840402, Tucson, Arizona
  - Investigational Site Number :840132, Little Rock, Arkansas
  - Investigational Site Number :840121, San Jose, California
  - Investigational Site Number :840403, Denver, Colorado
  - Investigational Site Number :840130, Denver, Colorado
  - Investigational Site Number :840115, Ocoee, Florida
  - Investigational Site Number :840055, Sarasota, Florida
  - Investigational Site Number :840079, Twin Falls, Idaho
  - Investigational Site Number :840032, Fort Mitchell, Kentucky
  - Investigational Site Number :840064, Bangor, Maine
  - Investigational Site Number :840052, Chevy Chase, Maryland
  - Investigational Site Number :840073, Gaithersburg, Maryland
  - Investigational Site Number :840018, Minneapolis, Minnesota
  - Investigational Site Number :840102, St Louis, Missouri
  - Investigational Site Number :840004, Papillion, Nebraska
  - Investigational Site Number :840068, West Long Branch, New Jersey
  - Investigational Site Number :840126, Charlotte, North Carolina
  - Investigational Site Number :840907, High Point, North Carolina
  - Investigational Site Number :840942, Toledo, Ohio
  - Investigational Site Number :840067, Philadelphia, Pennsylvania
  - Investigational Site Number :840091, Pittsburgh, Pennsylvania
  - Investigational Site Number :840070, Allen, Texas
  - Investigational Site Number :840062, Amarillo, Texas
  - Investigational Site Number :840124, Cypress, Texas
  - Investigational Site Number :840023, Dallas, Texas
  - Investigational Site Number :840922, Fort Worth, Texas
  - Investigational Site Number :840027, Fort Worth, Texas
  - Investigational Site Number :840008, San Antonio, Texas
  - Investigational Site Number :840035, Draper, Utah
  - Investigational Site Number :840077, Murray, Utah
  - Investigational Site Number :840057, South Burlington, Vermont
  - Investigational Site Number :840059, Fairfax, Virginia
  - Investigational Site Number :840951, Bellingham, Washington
- Argentina (12):
  - Investigational Site Number :032096, Bahía Blanca, Buenos Aires
  - Investigational Site Number :032091, Capital Federal, Buenos Aires
  - Investigational Site Number :032002, La Plata, Buenos Aires
  - Investigational Site Number :032006, Rosario, Santa Fe Province
  - Investigational Site Number :032005, Rosario, Santa Fe Province
  - Investigational Site Number :032004, Buenos Aires
  - Investigational Site Number :032003, Ciudad Autonoma Bs As
  - Investigational Site Number :032097, Ciudad Autonoma Buenos Aires
  - Investigational Site Number :032010, Ciudad Autonoma Buenos Aires
  - Investigational Site Number :032001, Ciudad Autonoma Buenos Aires
  - Investigational Site Number :032012, San Miguel de Tucumán
  - Investigational Site Number :032009, San Miguel de TucumÃ¡n
- Investigational Site Number :056003, Ghent, Belgium
- Canada (11):
  - Investigational Site Number :124006, Vancouver, British Columbia
  - Investigational Site Number :124017, Vancouver, British Columbia
  - Investigational Site Number :124016, Hamilton, Ontario
  - Investigational Site Number :124013, Ottawa, Ontario
  - Investigational Site Number :124002, Toronto, Ontario
  - Investigational Site Number :124010, MontrÃ©al, Quebec
  - Investigational Site Number :124001, Montreal, Quebec
  - Investigational Site Number :124012, Montreal, Quebec
  - Investigational Site Number :124014, QuÃ©bec, Quebec
  - Investigational Site Number :124007, Trois-Rivières, Quebec
  - Investigational Site Number :124018, Québec
- France (7):
  - Investigational Site Number :250009, Brest
  - Investigational Site Number :250010, Lille
  - Investigational Site Number :250006, Lyon
  - Investigational Site Number :250001, Marseille
  - Investigational Site Number :250002, Montpellier
  - Investigational Site Number :250005, Nantes
  - Investigational Site Number :250008, Strasbourg
- Germany (5):
  - Investigational Site Number :276006, Berlin
  - Investigational Site Number :276010, Frankfurt am Main
  - Investigational Site Number :276011, Großhansdorf
  - Investigational Site Number :276009, Koblenz
  - Investigational Site Number :276005, Rüdersdorf
- Israel (3):
  - Investigational Site Number :376001, Kfar Saba
  - Investigational Site Number :376005, Petah Tikva
  - Investigational Site Number :376002, Rehovot
- Japan (50):
  - Investigational Site Number :392106, Mizunami-shi, Gifu
  - Investigational Site Number :392043, Ota-shi, Gunma
  - Investigational Site Number :392021, Fukuyama-shi, Hiroshima
  - Investigational Site Number :392108, Hiroshima, Hiroshima
  - Investigational Site Number :392164, Muroran-shi, Hokkaido
  - Investigational Site Number :392008, Sapporo, Hokkaido
  - Investigational Site Number :392034, Sapporo, Hokkaido
  - Investigational Site Number :392006, Tomakomai-shi, Hokkaido
  - Investigational Site Number :392162, Kobe, Hyōgo
  - Investigational Site Number :392020, Naka-gun, Ibaraki
  - Investigational Site Number :392011, Sakaide-shi, Kagawa-ken
  - Investigational Site Number :392014, Yokohama, Kanagawa
  - Investigational Site Number :392153, Kyoto, Kyoto
  - Investigational Site Number :392170, Osaki-shi, Miyagi
  - Investigational Site Number :392045, Uruma, Okinawa
  - Investigational Site Number :392119, Kishiwada-shi, Osaka
  - Investigational Site Number :392005, Naruto-shi, Tokushima
  - Investigational Site Number :392002, Chuo-ku, Tokyo
  - Investigational Site Number :392112, Chuo-ku, Tokyo
  - Investigational Site Number :392133, Machida-shi, Tokyo
  - Investigational Site Number :392177, Ome-shi, Tokyo
  - Investigational Site Number :392038, Setagaya-ku, Tokyo
  - Investigational Site Number :392167, Shinagawa-ku, Tokyo
  - Investigational Site Number :392173, Tachikawa-shi, Tokyo
  - Investigational Site Number :392185, Akashi-shi
  - Investigational Site Number :392007, Chūōku
  - Investigational Site Number :392012, Edogawa-ku
  - Investigational Site Number :392030, Habikino-shi
  - Investigational Site Number :392004, Himeji-shi
  - Investigational Site Number :392158, Hiroshima
  - Investigational Site Number :392013, Iizuka-shi
  - Investigational Site Number :392042, Isesaki-shi
  - Investigational Site Number :392142, Kasuga-shi
  - Investigational Site Number :392040, Kodaira-shi
  - Investigational Site Number :392044, Kokubunji-shi
  - Investigational Site Number :392010, Kurashiki-shi
  - Investigational Site Number :392036, Kyoto
  - Investigational Site Number :392144, Minatoku
  - Investigational Site Number :392122, Minatoku
  - Investigational Site Number :392163, Nagoya
  - Investigational Site Number :392155, Osakasayama-shi
  - Investigational Site Number :392152, Osakasayama-shi
  - Investigational Site Number :392127, Ōta-ku
  - Investigational Site Number :392169, Sagamihara-shi
  - Investigational Site Number :392130, Shinjuku-ku
  - Investigational Site Number :392165, Sumida-ku
  - Investigational Site Number :392146, Tachikawa-shi
  - Investigational Site Number :392029, Tsu
  - Investigational Site Number :392168, Uozu-shi
  - Investigational Site Number :392132, Urasoe-shi
- Investigational Site Number :528001, Arnhem, Netherlands
- South Africa (7):
  - Investigational Site Number :710011, Cape Town
  - Investigational Site Number :710001, Cape Town
  - Investigational Site Number :710091, Cape Town
  - Investigational Site Number :710092, Cape Town
  - Investigational Site Number :710006, Durban
  - Investigational Site Number :710007, Pretoria
  - Investigational Site Number :710009, Winnie Mandela

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Maspero JF, Peters AT, Chapman KR, Domingo C, Stewart J, Hardin M, Maroni J, Tawo K, Khokhar FA, Mortensen E, Laws E, Radwan A, Jacob-Nara JA, Deniz Y, Rowe PJ. Long-Term Safety of Dupilumab in Patients With Moderate-to-Severe Asthma: TRAVERSE Continuation Study. J Allergy Clin Immunol Pract. 2024 Apr;12(4):991-997.e6. doi: 10.1016/j.jaip.2023.12.043. Epub 2023 Dec 30. PMID 38163585

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 138 sites in 10 countries. A total of 393 participants were enrolled in the study between 30 August 2018 and 27 August 2020.
Pre-assignment Details: Participants with moderate to severe asthma who had completed the parent study TRAVERSE-LTS12551 (NCT02134028) were enrolled in this current study (LPS15023).
Groups:
- Dupilumab: Participants received subcutaneous (SC) dose of dupilumab 300 milligrams (mg) every 2 weeks (q2w) from Week 0 up to Week 132. Participants who discontinued treatment for greater than or equal to [>=] 6 weeks after study LTS12551, received a 600 mg loading dose of dupilumab on Week 0. Participants were also on background dose of medium or high dose inhaled corticosteroid (ICS) as maintained in study LTS12551 in combination with controllers (and/or oral corticosteroid [OCS] for those participants from the original parent study EFC13691 [NCT02528214]). Salbutamol/albuterol hydrofluoroalkane pressurized metered dose inhalers (MDI) or levosalbutamol/levalbuterol hydrofluoroalkane pressurized MDI were given as reliever medication as needed during the study.
Period: Overall Study
Arm/Group | Dupilumab
Started | 393
Completed | 374
Not Completed | 19
Not completed — Participant decision | 7
Not completed — Adverse Event | 6
Not completed — Lack of Efficacy | 1
Not completed — Poor compliance to protocol | 2
Not completed — Other-unspecified | 3

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled participants.
Groups:
- Dupilumab: Participants received SC dose of dupilumab 300 mg q2w from Week 0 up to Week 132. Participants who discontinued treatment for >= 6 weeks after study LTS12551, received a 600 mg loading dose of dupilumab on Week 0. Participants were also on background dose of medium or high dose ICS as maintained in study LTS12551 in combination with controllers (and/or OCS for those participants from the original parent study EFC13691). Salbutamol/albuterol hydrofluoroalkane pressurized MDI or levosalbutamol/levalbuterol hydrofluoroalkane pressurized MDI were given as reliever medication as needed during the study.
Arm/Group | Dupilumab
Number analyzed (Participants) | 393
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (14.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 231
  Male | 162
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily had to have a causal relationship with the treatment. TEAEs were the AEs that developed or worsened or became serious during the TEAE period (defined as the time from the first dose of the investigational medicinal product [IMP] up to 12 weeks after the last dose of the IMP).
Time Frame: From first dose of IMP up to 12 weeks after last dose of IMP (maximum duration: up to 144 Weeks)
Population: Analysis was performed on safety population that included all participants who had actually received at least one dose or part of a dose of IMP.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 393
percentage of participants | 54.5 [47.40 to 62.26]

2. Primary Outcome: Treatment-emergent Adverse Event Rate (Event Per 100 Participant-years)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily had to have a causal relationship with the treatment. TEAEs were the AEs that developed or worsened or became serious during the TEAE period (defined as the time from the first dose of the IMP up to 12 weeks after last dose of the IMP). TEAE event rate was defined as the number of TEAE events per 100 participant-years.
Time Frame: From first dose of IMP up to 12 weeks after last dose of IMP (maximum duration: up to 144 Weeks)
Population: Analysis was performed on safety population.
Measure: Number (95% Confidence Interval); unit: events per 100 participant-years
Arm/Group | Dupilumab
Number analyzed (Participants) | 393
events per 100 participant-years | 171.4 [162.71 to 180.43]

3. Secondary Outcome: Adverse Events of Special Interest (AESIs) Event Rate (Event Per100 Participant-years)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily had to have a causal relationship with the treatment. AESIs were AE (serious or non-serious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the investigator to the Sponsor was required. AESI event rate was defined as the number of AESI events per 100 participant-years.
Time Frame: From first dose of IMP up to 12 weeks after last dose of IMP (maximum duration: up to 144 Weeks)
Population: Analysis was performed on safety population.
Measure: Number (95% Confidence Interval); unit: events per 100 participant-years
Arm/Group | Dupilumab
Number analyzed (Participants) | 393
events per 100 participant-years | 6.0 [4.40 to 7.99]

4. Secondary Outcome: Percentage of Participants With Treatment-emergent Serious Adverse Events (TESAEs), Adverse Events of Special Interest (AESIs) and AEs Leading to Study Discontinuation
Description: AE: any untoward medical occurrence in participants that received IMP and did not necessarily had to have causal relationship with treatment. TEAEs: AEs developed/worsened in grade/become serious during the TEAE period (from first dose of IMP up to 12 weeks after last dose of IMP).SAE: any untoward medical occurrence at any dose resulted in death, was life-threatening, required inpatient hospitalization, prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was congenital anomaly/birth defect or was medically important event. AESI: AE (serious/non-serious) of scientific and medical concern specific to Sponsor's product/program, for which ongoing monitoring and immediate notification by Investigator to Sponsor required.
Time Frame: From first dose of IMP up to 12 weeks after last dose of IMP (maximum duration: up to 144 Weeks)
Population: Analysis was performed on safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 393
percentage of participants
  TESAEs | 5.6
  AESIs | 6.1
  AEs leading to study discontinuation | 1.5

ADVERSE EVENTS:
Time Frame: From first dose of IMP up to 12 weeks after last dose of IMP (maximum duration: up to 144 Weeks)
Description: Reported AEs and deaths were TEAEs that developed or worsened or became serious during the TEAE period (defined as the time from the first dose of the IMP up to 12 weeks after last dose of the IMP). Analysis was performed on safety population.
Arm/Group | Dupilumab
All-Cause Mortality (participants affected / at risk) | 5/393
Serious Adverse Events (participants affected / at risk) | 22/393
Other Adverse Events (participants affected / at risk) | 93/393
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab (N=393)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Pudendal canal syndrome (Nervous system disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab (N=393)
Asthma (Respiratory, thoracic and mediastinal disorders) | 52 (77)
COVID-19 (Infections and infestations) | 22 (24)
Nasopharyngitis (Infections and infestations) | 33 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT03620747/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT03620747/SAP_001.pdf